CLINICAL TRIAL: NCT01067833
Title: A Pilot Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multi-Centered Safety, Tolerability and Preliminary EffiCacy Study of K201 Oral for the Prevention of ATrial FIbrillation (AF) Recurrence in Subjects Post-Conversion From AF
Brief Title: Phase 2 Study of Oral K201 for Prevention of AF Recurrence
Acronym: ARCTIC-AF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sequel Pharmaceuticals, Inc (Industry)
Responsible Party: Howard C. Dittrich, CMO, Sequel Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CJO-201
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; AF
MeSH Terms: conditions — Atrial Fibrillation | interventions — K201 compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Tablet
- Dose 1 (Experimental): K201
  Interventions: Drug: K201 Tablet
- Dose 2 (Experimental): K201
  Interventions: Drug: K201 Tablet
- Dose 3 (Experimental): K201
  Interventions: Drug: K201 Tablet

INTERVENTIONS:
Drug: K201 Tablet — oral tablet, x28 days
  Arms: Dose 1; Dose 2; Dose 3
Drug: Placebo Tablet — oral tablet, x28 days
  Arms: Placebo

SUMMARY:
To evaluate the safety, efficacy, and tolerability of 3 doses of K201 (oral) administered for up to 28 days in subjects with recent DC cardioversion to sinus rhythm from sustained symptomatic atrial fibrillation (AF duration >3 days and <6 months).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic AF (sustained >3 days and <6 months) and clinically indicated for cardioversion;
* Adequate anticoagulant therapy for cardioversion in accordance with standard practice as recommended by ACC/AHA/ESC guidelines or with local clinical practice;
* Hemodynamically stable (90 mmHg < systolic blood pressure < 190 mmHg)at screening and on Day 1;

Exclusion Criteria:

* Known prolonged QT syndrome or QTc interval of >0.500 sec at screening; familial long QT syndrome; previous Torsade de Pointes; ventricular fibrillation; or sustained ventricular tachycardia (VT);
* QRS >0.130 sec;
* Previous episodes of second- or third-degree atrioventricular block;
* Unsuccessful DC cardioversion attempt within 3 months; prior ablation for AF;
* Persistent bradycardia with ventricular rate below 50 beats/min, sick-sinus syndrome or pacemaker (including CRT, AICD);
* Myocardial infarction (MI), cardiac surgery, angioplasty, unstable angina or acute coronary syndrome within 30 days prior to entry into the study;
* NYHA Class III or Class IV heart failure (HF) at screening or admission, or hospitalized for HF in previous 6 months;
* Known concurrent temporary secondary causes of AF;
* Received a Class I or Class III antiarrhythmic agent (including sotalol) within 5 half-lives of randomization or amiodarone or dronedarone within 4 weeks;
* Received treatment with other drugs known to prolong the QT interval within 5 half-lives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
time to first documented recurrence of symptomatic AF | 28 days
time to first documented recurrence of symptomatic or asymptomatic AF | 28 days
proportion of subjects in sinus rhythm | Day 28
number of AF beats | 10 days
time in AF | 10 days
safety assessments: vital signs, laboratory assays, ECG parameters, physical exams, frequency of adverse events | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chamberlin, MD, Study Director — Sequel Pharmaceuticals